CLINICAL TRIAL: NCT04798573
Title: Phenomics and Genomics of Clinically Relevant Chronic Postsurgical Pain: A Multicenter Prospective Study
Brief Title: Phenomics and Genomics of Clinically Relevant Chronic Postsurgical Pain
Acronym: CT-Pain
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 12-0078
Record Dates: First submitted 2021-01-07; First posted 2021-03-15 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain; Surgery
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will extract DNA from blood and contrast the genetic variations of participants with clinically significant chronic pain, to identify variations associated with the development of chronic post-surgical pain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The investigators will approach elective cardiac and thoracic surgery patients in the preoperative consultation clinic. Consenting individuals will be administered, before surgery validated pain, psychological and sleep questionnaires. These questionnaires will be repeated at 3, 6 and 12 months postoperatively (PO) to follow up the progression of early PO pain and the transition to chronicity. Participants will define clinically relevant pain by calculating a chronic pain index (CPI). In addition, the investigators will follow the development of acute postsurgical and chronic pain from before surgery up to a year after, extract DNA from blood and contrast the genetic variations of participants with clinically significant chronic pain, to identify variations associated with the development of chronic post-surgical pain.

DETAILED DESCRIPTION:
Most patients who undergo surgery heal within weeks to months and return to their baseline functional status or to an improved level of functioning. However, some patients have pain after surgery which continues. The purpose of this study is to see if there is a relationship between patient's genetic makeup (diseases that are passed on in families) and pain experience following cardiac and thoracic surgeries. This study will look for links between psychological factors, environmental factors and genetic factors in an attempt to uncover the risk for developing chronic post-surgical pain.

This study hopes to determine differences between traditional pain surveys and a basic science approach called "Phenomics" to measure chronic pain response after cardiac and thoracic surgery. Phenomics or Phenomes is the study of physical characteristics, outside influences and biochemical changes (traits or chemical characteristics) and their response to either the environment or genetic changes. Validated pain questionnaires will be administered before surgery, and will repeated at 3, 6, and 12 months postoperatively to follow up the progression of early postoperative pain and the transition to chronicity. In general, the psychological and pain questionnaires are designed to measure the following: anxiety, thoughts, feelings and reactions toward pain and stressful experiences.

In addition, the study will follow the development of acute postoperative and chronic pain from before surgery up to a year after. The investigators will extract DNA from blood and contrast the genetic variations of participants with clinically significant chronic pain, to identify variations associated with the development of chronic post-surgical pain. The blood sample will be drawn at the time of the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Non- Emergency Cardiac Surgery with Midline Sternotomy OR Thoracic Surgery via VATS or Lateral Thoracotomy
3. Written informed consent to participate in the study

Exclusion Criteria:

1. Patient unable to understand the study protocol
2. History of a psychotic psychiatric disorder
3. Unable to speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective cardiac and thoracic surgery patients who agree to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2012-08-03 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Post-Surgical Pain Intensity | 1 year from the day of surgery
  Measured using the numeric rating scale (0=no pain; 10=worst pain imaginable)
Pain: Measured using the McGill Pain Questionnaire- Short Form-2 (SF-MPQ-2) | 1 year from the day of surgery
  The SF-MPQ-2 is a 22-item, expanded and revised version of the SF-MPQ designed to measure the qualities of neuropathic and non-neuropathic pain. Exploratory and confirmatory factor analyses revealed the presence of the following four factors or subscales: (1) continuous pain, (2) intermittent pain, (3) neuropathic pain, and (4) affective pain descriptor.
Pain: Measured using the Self-completed Leeds Assessment of Neuropathic Symptoms and Signs (SLANSS) | 1 year from the day of surgery
  The S-LANSS is a validated 7-item questionnaire designed to distinguish whether pain is predominately neuropathic or nociceptive in origin.
Anxiety: Measured using the Anxiety Sensitivity Index-3 (ASI-3) | 1 year from the day of surgery
  The ASI-3 is a revised version of the widely used, 16-item scale ASI that measures concerns that anxiety and anxiety-related symptoms will lead to harmful negative consequences. Each item is rated on a 5-point scale ranging from very little (0) to very much (4).
Pain Catastrophizing: Measured using the Pain Catastrophizing Scale (PCS) | 1 year from the day of surgery
  The PCS consists of 13 items describing thoughts and feelings that individuals may experience when they are in pain. Each item is rated on a 5-point scale ranging from not at all (0) to all the time (4).
Pain Anxiety: Measured using the Pain Anxiety Symptoms Scale-20 (PASS-20) | 1 year from the day of surgery
  The PASS-20 is a shortened 20-item version of the original Pain Anxiety Symptoms Scale designed to measure fear and anxiety responses specific to pain, including avoidance. The PASS-20 has four 5-item subscales, including (1) cognitive anxiety, (2) escape and avoidance, (3) fearful thinking, and (4) physiological anxiety.
Pain Disability: Measured using the Pain Disability Index (PDI) | 1 year from the day of surgery
  The PDI assesses the extent to which persistent pain interferes with an individual's ability to engage in seven different areas of everyday activity including: (1) family/home responsibilities, (2) recreation, (3) social activity, (4) occupation, (5) sexual behavior, (6) self-care, and (7) life-support activity.
Posttraumatic Stress Disorder: Measured using the Posttraumatic Stress Disorder Checklist-Civilian Version (PCL-C) | 1 year from the day of surgery
  The Posttraumatic Stress Disorder Checklist - Civilian Version (PCL-C) is a 17-item self-report measure based on the current DSM-IV symptoms for PTSD. Respondents are asked to indicate how much they have been bothered by each symptom 5-point scale ranging from not at all (1) to extremely (5).
Anxiety and Depression: Measured using The Hospital Anxiety and Depression Scale (HADS) | 1 year from the day of surgery
  The HADS is the most widely used scale for measuring symptoms of anxiety and depression among medical inpatients, outpatients and the general population and consists of 7 anxiety and 7 depression-related items.
Somatization: Measured using the SCL-90-R-Somatization | 1 year from the day of surgery
  The SCL-90-R is a widely-used self-report symptom inventory measuring psychological symptoms of psychiatric and medical patients. Participants rate each item on a five-point scale of distress, ranging from 0 (no distress) to 4 (extreme distress).
Chronic Pain Acceptance: Measured using the Chronic Pain Acceptance Questionnaire (CPAQ) | 1 year from the day of surgery
  The CPAQ is a 20-item questionnaire that measures how participants react and adapt to living with chronic pain. Participants respond to "how true" each item is by selecting a number from 0 ("never true") to 6 ("always true").
Mindful Attention Awareness: Measured using the Mindful Attention Awareness Scale (MAAS) | 1 year from the day of surgery
  The MAAS is a 15-item scale designed to measure a central feature of dispositional mindfulness characterized by "open or receptive awareness of and attention to" the present. Participants respond to how frequently/infrequently they experience each item by selecting one of six response options on a Likert rating scale ranging from 1 ("Almost always") to 6 ("Almost never").
Pain Self Efficacy: Measured using the Pain Self-Efficacy Questionnaire (PSEQ) | 1 year from the day of surgery
  The PSEQ is a 10-item Likert-type questionnaire, designed specifically for chronic pain, where patients are asked to rate their confidence to complete certain activities despite pain.
Sensitivity to Pain Traumatization: Measured using the Sensitivity to Pain Traumatization Scale (SPTS) | 1 year from the day of surgery
  The SPTS is a 12-item questionnaire that was designed to measure the anxiety-related cognitive, emotional and behavioural reactions to pain that resemble symptoms of a traumatic stress reaction. Each item is rated on a 5-item Likert scale (from 1 (not at all true) to 5 (entirely true)).
Sleep Problems: Measured using the Sleep Problems Questionnaire | 1 year from the day of surgery
  This is a general questionnaire that asks its questions providing responses in units of days.
Sleep Quality: Measured using the Pittsburg Sleep Quality Index (PQSI) | 1 year from the day of surgery
  The PSQI questionnaire is much more specific, identifying specific responses and reasons why patients may be having trouble sleeping such as: (1) cannot get to sleep within 30 minutes and (2) wake up in the middle of the night or early morning.

SECONDARY OUTCOMES:
Physical Activity for Thoracic Patients: Measured using Actiwatch--64 | Up to 11 days from surgery
  The Actiwatch-64 is a small wrist watch-like device that contains an accelerometer that records limb movements and has a memory storage capacity for up to 11 days109. The Actiwatch-64 provides a non-invasive method of collecting activity data around the clock. Activity data are downloaded to a laptop and standard sleep parameters such as latency to sleep (SOL), wake time after sleep onset (WASO), and total sleep time (TST) are inferred by software based on the presence and absence of limb movements during specified time intervals. Total activity during periods scored as not sleep is also available.
Sleep Quality for Thoracic Patients: Measured using the Sleep Quality Assessment | Up to 11 days from surgery
  Each morning after surgery, up to and including the morning of discharge home from the hospital, a Sleep Diary will be completed.
Mechanical Pain Pressure: Measured using the Mechanical Pressure Pain Threshold (PPT) | 1 year from the day of surgery
  Pain thresholds in response to mechanical pressure applied to the skin will be obtained using a Pressure Algometer.
Thermal Pain and Sensory: Measured using the Thermal Pain and Sensory Thresholds | 1 year from the day of surgery
  Thermal stimuli will be delivered using the Medoc Thermal NeuroSensory Analyzer
Pain Illusion: Measured using the Thermal Grill Illusion Test | 1 year from the day of surgery
  Participants will be required to place their right hand on four plates, two of which will be pre-cooled to 10˚C and 20˚C and two preheated to 40˚C and 50˚C. Participants will alternate between these stimuli and a grill of mixed 20˚C and 40˚C interlaced bars with 5sec intervals between applications.
Pain: Measured using the Vasoconstrictor Inspiratory Gasp | 1 year from the day of surgery
  This simple test robustly activates the sympathetic system, which aggravates neuropathic pain in some chronic pain patients. Participants will be asked to rest supine on a couch and relax with eyes closed, and to take the deepest possible inspiration and then breathe normally. Three ratings of ongoing spontaneous pain will be taken at 1, 2, and 5 min after expiration. Two baseline blood pressure (systolic, diastolic and mean arterial pressure) and pulse rate measurements will be taken just before the Gasp Test and at 1 and 2 min thereafter, just after the pain ratings. Cardiovascular parameters will be carried out using an automated blood pressure cuff.
Cold Pressor Pain: Measured using the Cold Pressor Pain Test | 1 year from the day of surgery
  The participant will immerse their right hand (above the elbow) in ice cold water and keep it there until they cannot tolerate the pain. The pain tolerance threshold will be recorded with a stopwatch, as the time to withdrawal; cut-off at 3 min. They will then use the NRS (0-100) to rate the magnitude of pain and unpleasantness.

OTHER OUTCOMES:
Genotyping Outcomes- DNA and Biomarkers | From pre-surgery to 3 month post-surgically
  A genome-wide exomic sequencing and full genome sequencing will be carried out in search of a common and rare variants that predispose carriers to acute post-surgical pain and the transition to pain chronicity post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hance Clarke, MD PhD FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohayon MM, Schatzberg AF. Chronic pain and major depressive disorder in the general population. J Psychiatr Res. 2010 May;44(7):454-61. doi: 10.1016/j.jpsychires.2009.10.013. Epub 2010 Feb 9. PMID 20149391
- [Background] Wall PD, Jones M. Defeating pain: The war against a silent epidemic. New York, NY: Plenum Press; 1991.
- [Background] McCarberg BH, Billington R. Consequences of neuropathic pain: quality-of-life issues and associated costs. Am J Manag Care. 2006 Jun;12(9 Suppl):S263-8. PMID 16774458
- [Background] Diatchenko L, Slade GD, Nackley AG, Bhalang K, Sigurdsson A, Belfer I, Goldman D, Xu K, Shabalina SA, Shagin D, Max MB, Makarov SS, Maixner W. Genetic basis for individual variations in pain perception and the development of a chronic pain condition. Hum Mol Genet. 2005 Jan 1;14(1):135-43. doi: 10.1093/hmg/ddi013. Epub 2004 Nov 10. PMID 15537663
- [Background] Katz J, Seltzer Z. Transition from acute to chronic postsurgical pain: risk factors and protective factors. Expert Rev Neurother. 2009 May;9(5):723-44. doi: 10.1586/ern.09.20. PMID 19402781
- [Background] Max MB, Stewart WF. The molecular epidemiology of pain: a new discipline for drug discovery. Nat Rev Drug Discov. 2008 Aug;7(8):647-58. doi: 10.1038/nrd2595. Epub 2008 Jun 27. PMID 18587382
- [Background] Seltzer Z, Dorfman R. Identifying genetic and environmental risk factors for chronic orofacial pain syndromes: human models. J Orofac Pain. 2004 Fall;18(4):311-7. PMID 15636014
- [Background] Seltzer Z, Mogil JS. Pain and genetics. In: Sessle BJ, Lavigne GJ, Lund JP, Dubner R (eds). Orofacial Pain and Related Conditions. 2nd edition ed. Hanover Park, Illinois: Quintessence Publishing, 2008:69-75.
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Crombie IK, Davies HT, Macrae WA. Cut and thrust: antecedent surgery and trauma among patients attending a chronic pain clinic. Pain. 1998 May;76(1-2):167-71. PMID 9696470
- [Background] King KM, Tsuyuki R, Faris P, Currie G, Maitland A, Collins-Nakai RL. A randomized controlled trial of women's early use of a novel undergarment following sternotomy: the Women's Recovery from Sternotomy Trial (WREST). Am Heart J. 2006 Dec;152(6):1187-93. doi: 10.1016/j.ahj.2006.07.026. PMID 17161074
- [Background] King KM, Parry M, Southern D, Faris P, Tsuyuki RT. Women's Recovery from Sternotomy-Extension (WREST-E) study: examining long-term pain and discomfort following sternotomy and their predictors. Heart. 2008 Apr;94(4):493-7. doi: 10.1136/hrt.2007.117606. Epub 2007 Jul 16. PMID 17639091
- [Background] Lahtinen P, Kokki H, Hynynen M. Pain after cardiac surgery: a prospective cohort study of 1-year incidence and intensity. Anesthesiology. 2006 Oct;105(4):794-800. doi: 10.1097/00000542-200610000-00026. PMID 17006079
- [Background] Meyerson J, Thelin S, Gordh T, Karlsten R. The incidence of chronic post-sternotomy pain after cardiac surgery--a prospective study. Acta Anaesthesiol Scand. 2001 Sep;45(8):940-4. doi: 10.1034/j.1399-6576.2001.450804.x. PMID 11576043
- [Background] Routledge FS, Tsuyuki RT, Hervas-Malo M, LeBlanc P, McFetridge-Durdle JA, King KM. The influence of coronary artery bypass graft harvest site on women's pain, functional status, and health services utilization throughout the first post-operative year: a longitudinal study. Int J Nurs Stud. 2009 Aug;46(8):1054-60. doi: 10.1016/j.ijnurstu.2009.02.003. Epub 2009 Mar 9. PMID 19269633
- [Background] Lopez V, Sek Ying C, Poon CY, Wai Y. Physical, psychological and social recovery patterns after coronary artery bypass graft surgery: a prospective repeated measures questionnaire survey. Int J Nurs Stud. 2007 Nov;44(8):1304-15. doi: 10.1016/j.ijnurstu.2006.06.005. Epub 2006 Aug 30. PMID 16942769
- [Background] Gjeilo KH, Stenseth R, Wahba A, Lydersen S, Klepstad P. Validation of the brief pain inventory in patients six months after cardiac surgery. J Pain Symptom Manage. 2007 Dec;34(6):648-56. doi: 10.1016/j.jpainsymman.2007.01.010. Epub 2007 Jul 16. PMID 17629665
- [Background] Wildgaard K, Ravn J, Nikolajsen L, Jakobsen E, Jensen TS, Kehlet H. Consequences of persistent pain after lung cancer surgery: a nationwide questionnaire study. Acta Anaesthesiol Scand. 2011 Jan;55(1):60-8. doi: 10.1111/j.1399-6576.2010.02357.x. Epub 2010 Nov 15. PMID 21077845
- [Background] Kristensen AD, Pedersen TA, Hjortdal VE, Jensen TS, Nikolajsen L. Chronic pain in adults after thoracotomy in childhood or youth. Br J Anaesth. 2010 Jan;104(1):75-9. doi: 10.1093/bja/aep317. PMID 19915188
- [Background] Steegers MA, Snik DM, Verhagen AF, van der Drift MA, Wilder-Smith OH. Only half of the chronic pain after thoracic surgery shows a neuropathic component. J Pain. 2008 Oct;9(10):955-61. doi: 10.1016/j.jpain.2008.05.009. Epub 2008 Jul 16. PMID 18632308
- [Background] Maguire MF, Ravenscroft A, Beggs D, Duffy JP. A questionnaire study investigating the prevalence of the neuropathic component of chronic pain after thoracic surgery. Eur J Cardiothorac Surg. 2006 May;29(5):800-5. doi: 10.1016/j.ejcts.2006.02.002. Epub 2006 Apr 3. PMID 16581259
- [Background] Kalso E, Perttunen K, Kaasinen S. Pain after thoracic surgery. Acta Anaesthesiol Scand. 1992 Jan;36(1):96-100. doi: 10.1111/j.1399-6576.1992.tb03430.x. PMID 1539485
- [Background] Bruce J, Drury N, Poobalan AS, Jeffrey RR, Smith WC, Chambers WA. The prevalence of chronic chest and leg pain following cardiac surgery: a historical cohort study. Pain. 2003 Jul;104(1-2):265-73. doi: 10.1016/s0304-3959(03)00017-4. PMID 12855337
- [Background] Eisenberg E, Pultorak Y, Pud D, Bar-El Y. Prevalence and characteristics of post coronary artery bypass graft surgery pain (PCP). Pain. 2001 May;92(1-2):11-7. doi: 10.1016/s0304-3959(00)00466-8. PMID 11323122
- [Background] Kalso E, Mennander S, Tasmuth T, Nilsson E. Chronic post-sternotomy pain. Acta Anaesthesiol Scand. 2001 Sep;45(8):935-9. doi: 10.1034/j.1399-6576.2001.450803.x. PMID 11576042
- [Background] Steegers MA, van de Luijtgaarden A, Noyez L, Scheffer GJ, Wilder-Smith OH. The role of angina pectoris in chronic pain after coronary artery bypass graft surgery. J Pain. 2007 Aug;8(8):667-73. doi: 10.1016/j.jpain.2007.04.007. Epub 2007 Jun 13. PMID 17569594
- [Background] Searle RD, Simpson MP, Simpson KH, Milton R, Bennett MI. Can chronic neuropathic pain following thoracic surgery be predicted during the postoperative period? Interact Cardiovasc Thorac Surg. 2009 Dec;9(6):999-1002. doi: 10.1510/icvts.2009.216887. Epub 2009 Sep 18. PMID 19767301
- [Background] Katz J, Asmundson GJ, McRae K, Halket E. Emotional numbing and pain intensity predict the development of pain disability up to one year after lateral thoracotomy. Eur J Pain. 2009 Sep;13(8):870-8. doi: 10.1016/j.ejpain.2008.10.003. Epub 2008 Nov 21. PMID 19027333
- [Background] Gottschalk A, Ochroch EA. Clinical and demographic characteristics of patients with chronic pain after major thoracotomy. Clin J Pain. 2008 Oct;24(8):708-16. doi: 10.1097/AJP.0b013e318174badd. PMID 18806536
- [Background] Senturk M, Ozcan PE, Talu GK, Kiyan E, Camci E, Ozyalcin S, Dilege S, Pembeci K. The effects of three different analgesia techniques on long-term postthoracotomy pain. Anesth Analg. 2002 Jan;94(1):11-5, table of contents. doi: 10.1213/00000539-200201000-00003. PMID 11772793
- [Background] Guastella V, Mick G, Soriano C, Vallet L, Escande G, Dubray C, Eschalier A. A prospective study of neuropathic pain induced by thoracotomy: incidence, clinical description, and diagnosis. Pain. 2011 Jan;152(1):74-81. doi: 10.1016/j.pain.2010.09.004. Epub 2010 Nov 13. PMID 21075523
- [Background] Gjeilo KH, Klepstad P, Wahba A, Lydersen S, Stenseth R. Chronic pain after cardiac surgery: a prospective study. Acta Anaesthesiol Scand. 2010 Jan;54(1):70-8. doi: 10.1111/j.1399-6576.2009.02097.x. Epub 2009 Aug 13. PMID 19681771
- [Background] Choinière M, Watt-Watson J, Costello J, Guerriere D, Carrier M, Cogan M, Bussieres J, Guertin MC, Lespérance F, Basket R, McFetridge-Durdle J, Sullivan J. Prevalence, characterictics, and risk factors of persistent post-operative pain after cardiac surgery. Pain Research and Management. 2009;14(2):144.
- [Background] Katz J. Pain begets pain - Predictors of long-term phantom limb pain and post-thoracotomy pain. Pain Forum. 1997;6:140-4.
- [Background] Katz J, Jackson M, Kavanagh BP, Sandler AN. Acute pain after thoracic surgery predicts long-term post-thoracotomy pain. Clin J Pain. 1996 Mar;12(1):50-5. doi: 10.1097/00002508-199603000-00009. PMID 8722735
- [Background] Kidd BL, Urban LA. Mechanisms of inflammatory pain. Br J Anaesth. 2001 Jul;87(1):3-11. doi: 10.1093/bja/87.1.3. No abstract available. PMID 11460811
- [Background] Tajerian M, Clark JD. The role of the extracellular matrix in chronic pain following injury. Pain. 2015 Mar;156(3):366-370. doi: 10.1097/01.j.pain.0000460323.80020.9d. No abstract available. PMID 25679468
- [Background] Kim H, Ramsay E, Lee H, Wahl S, Dionne RA. Genome-wide association study of acute post-surgical pain in humans. Pharmacogenomics. 2009 Feb;10(2):171-9. doi: 10.2217/14622416.10.2.171. PMID 19207018
- [Background] Lu Y, Belfer I, Vatine JJ, Shir Y, Jablonski-Peetz T, Pfeffer RM, Hipp H, Sun L, Craiu R, Goldman D, Max MB, Seltzer Z. Neuropathic pain levels following surgical nerve injury are controlled by genotypes and haplotypes of COMT - the gene encoding catecholamine-o-methyltransferase.Second International Conference on Neuropathic Pain. Berlin, Germany, 2007.
- [Background] Lu Y, Belfer I, Gershon E, Vatine JJ, Shir Y, Jablonski-Peetz T, Pfeffer RM, Hipp H, Livneh J, Goldman D, Max M, Seltzer Z. Do GCH1 polymorphisms control the risk for developing chronic pain in leg amputees and women postmastectomy? . Canadian Association of Genetic Epidemiology. Toronto, Canada, 2007.
- [Background] Seltzer Z. Studying candidate genes for chronic pain: the example of COMT, the gene encoding Catechol-O-methyltransferase. 5th Congress of the European Federation of IASP Chapters (EFIC). Istanbul, Turkey 2006:13-6.
- [Background] Nissenbaum J, Devor M, Seltzer Z, Gebauer M, Michaelis M, Tal M, Dorfman R, Abitbul-Yarkoni M, Lu Y, Elahipanah T, delCanho S, Minert A, Fried K, Persson AK, Shpigler H, Shabo E, Yakir B, Pisante A, Darvasi A. Susceptibility to chronic pain following nerve injury is genetically affected by CACNG2. Genome Res. 2010 Sep;20(9):1180-90. doi: 10.1101/gr.104976.110. Epub 2010 Aug 5. PMID 20688780
- [Background] Costigan M, Belfer I, Griffin RS, Dai F, Barrett LB, Coppola G, Wu T, Kiselycznyk C, Poddar M, Lu Y, Diatchenko L, Smith S, Cobos EJ, Zaykin D, Allchorne A, Gershon E, Livneh J, Shen PH, Nikolajsen L, Karppinen J, Mannikko M, Kelempisioti A, Goldman D, Maixner W, Geschwind DH, Max MB, Seltzer Z, Woolf CJ. Multiple chronic pain states are associated with a common amino acid-changing allele in KCNS1. Brain. 2010 Sep;133(9):2519-27. doi: 10.1093/brain/awq195. Epub 2010 Aug 18. PMID 20724292
- [Background] Sackstein M, Ramer A, Seltzer Z. Specific patterns of injury discharge are associated with receptor types in freshly injured sensory myelinated (A-) and unmyelinated (C-) fibers in rat. 8th World Congress on Pain. Vancouver, Canada, 1996.
- [Background] Seltzer Z, Beilin B, Ginzburg R, Paran Y, Shimko T. The role of injury discharge in the induction of neuropathic pain behavior in rats. Pain. 1991 Sep;46(3):327-336. doi: 10.1016/0304-3959(91)90115-E. PMID 1758712
- [Background] Seltzer Z, Cohn S, Ginzburg R, Beilin B. Modulation of neuropathic pain behavior in rats by spinal disinhibition and NMDA receptor blockade of injury discharge. Pain. 1991 Apr;45(1):69-75. doi: 10.1016/0304-3959(91)90166-U. PMID 1677750
- [Background] Cohn S, Seltzer Z. Inherited propensity for neuropathic pain is mediated by sensitivity to injury discharge. Neuroreport. 1991 Nov;2(11):647-50. doi: 10.1097/00001756-199111000-00003. PMID 1810457
- [Background] Sabsovich I, Neumann R, Dorfman J, Storm-Mathisen OP, Otterson P, Raber R, Zeltser R, Cevor M, Seltzer Z. Spinal dorsal horn inhibitory amino acid neurons: genetic differences and response to peripheral neurectomy. 3rd Congress of the European Federation of IASP Chapters (EFIC). Nice, France, 2000.
- [Background] Zhang SH, Blech-Hermoni Y, Faravelli L, Seltzer Z. Ralfinamide administered orally before hindpaw neurectomy or postoperatively provided long-lasting suppression of spontaneous neuropathic pain-related behavior in the rat. Pain. 2008 Oct 15;139(2):293-305. doi: 10.1016/j.pain.2008.04.020. Epub 2008 Jun 25. PMID 18583049
- [Background] Katz J, Clarke H. Preventive analgesia and beyond: Current status, evidence, and future directions. In: Macintyre PE, Rowbotham DJ, Howard R (eds). Clinical pain management: Acute pain 2nd ed. London: Hodder Arnold Ltd, 2008:154-98.
- [Background] McCartney CJ, Sinha A, Katz J. A qualitative systematic review of the role of N-methyl-D-aspartate receptor antagonists in preventive analgesia. Anesth Analg. 2004 May;98(5):1385-400, table of contents. doi: 10.1213/01.ane.0000108501.57073.38. PMID 15105220
- [Background] Katz J, Schmid R, Snijdelaar DG, Coderre TJ, McCartney CJL, Wowk A. Pre-emptive analgesia using intravenous fentanyl plus low-dose ketamine for radical prostatectomy under general anesthesia does not produce short-term or long-term reductions in pain or analgesic use. Pain. 2004 Aug;110(3):707-718. doi: 10.1016/j.pain.2004.05.011. PMID 15288412
- [Background] Clarke H, Pereira S, Kennedy D, Andrion J, Mitsakakis N, Gollish J, Katz J, Kay J. Adding gabapentin to a multimodal regimen does not reduce acute pain, opioid consumption or chronic pain after total hip arthroplasty. Acta Anaesthesiol Scand. 2009 Sep;53(8):1073-83. doi: 10.1111/j.1399-6576.2009.02039.x. Epub 2009 Jun 30. PMID 19572933
- [Background] Clarke H, Pereira S, Kennedy D, Gilron I, Katz J, Gollish J, Kay J. Gabapentin decreases morphine consumption and improves functional recovery following total knee arthroplasty. Pain Res Manag. 2009 May-Jun;14(3):217-22. doi: 10.1155/2009/930609. PMID 19547761
- [Background] Snijdelaar DG, Cornelisse HB, Schmid RL, Katz J. A randomised, controlled study of peri-operative low dose s(+)-ketamine in combination with postoperative patient-controlled s(+)-ketamine and morphine after radical prostatectomy. Anaesthesia. 2004 Mar;59(3):222-8. doi: 10.1111/j.1365-2044.2003.03620.x. PMID 14984518
- [Background] Snijdelaar DG, Koren G, Katz J. Effects of perioperative oral amantadine on postoperative pain and morphine consumption in patients after radical prostatectomy: results of a preliminary study. Anesthesiology. 2004 Jan;100(1):134-41. doi: 10.1097/00000542-200401000-00022. PMID 14695734
- [Background] Katz J, Clarke H, Seltzer Z. Review article: Preventive analgesia: quo vadimus? Anesth Analg. 2011 Nov;113(5):1242-53. doi: 10.1213/ANE.0b013e31822c9a59. Epub 2011 Sep 30. PMID 21965352
- [Background] Novak CB, Anastakis DJ, Beaton DE, Katz J. Patient-reported outcome after peripheral nerve injury. J Hand Surg Am. 2009 Feb;34(2):281-7. doi: 10.1016/j.jhsa.2008.11.017. PMID 19181228
- [Background] Gibas AL, Klatt R, Johnson J, Clarke JT, Katz J. A survey of the pain experienced by males and females with Fabry disease. Pain Res Manag. 2006 Autumn;11(3):185-92. doi: 10.1155/2006/828964. PMID 16960635
- [Background] Cohen L, Fouladi RT, Katz J. Preoperative coping strategies and distress predict postoperative pain and morphine consumption in women undergoing abdominal gynecologic surgery. J Psychosom Res. 2005 Feb;58(2):201-9. doi: 10.1016/j.jpsychores.2004.07.007. PMID 15820849
- [Background] Martin AL, Halket E, Asmundson GJ, Flora DB, Katz J. Posttraumatic stress symptoms and the diathesis-stress model of chronic pain and disability in patients undergoing major surgery. Clin J Pain. 2010 Jul-Aug;26(6):518-27. doi: 10.1097/AJP.0b013e3181e15b98. PMID 20551727
- [Background] Bar-El Y, Gilboa B, Unger N, Pud D, Eisenberg E. Skeletonized versus pedicled internal mammary artery: impact of surgical technique on post CABG surgery pain. Eur J Cardiothorac Surg. 2005 Jun;27(6):1065-9. doi: 10.1016/j.ejcts.2005.02.016. Epub 2005 Apr 8. PMID 15896618
- [Background] Edwards PW, Zeichner A, Kuczmierczyk AR, Boczkowski J. Familial pain models: the relationship between family history of pain and current pain experience. Pain. 1985 Apr;21(4):379-384. doi: 10.1016/0304-3959(85)90166-6. PMID 4000687
- [Background] Kusumi M, Araki H, Ijiri T, Kowa H, Adachi Y, Takeshima T, Sakai F, Nakashima K. Serotonin 2C receptor gene Cys23Ser polymorphism: a candidate genetic risk factor of migraine with aura in Japanese population. Acta Neurol Scand. 2004 Jun;109(6):407-9. doi: 10.1111/j.1600-0404.2004.00236.x. PMID 15147464
- [Background] Borroni B, Brambilla C, Liberini P, Rao R, Archetti S, Gipponi S, Volta GD, Padovani A. Functional serotonin 5-HTTLPR polymorphism is a risk factor for migraine with aura. J Headache Pain. 2005 Sep;6(4):182-4. doi: 10.1007/s10194-005-0179-9. PMID 16362658
- [Background] Guimaraes AL, de Sa AR, Victoria JM, de Fatima Correia-Silva J, Gomez MV, Gomez RS. Interleukin-1beta and serotonin transporter gene polymorphisms in burning mouth syndrome patients. J Pain. 2006 Sep;7(9):654-8. doi: 10.1016/j.jpain.2006.02.011. PMID 16942951
- [Background] Camilleri M, Busciglio I, Carlson P, McKinzie S, Burton D, Baxter K, Ryks M, Zinsmeister AR. Candidate genes and sensory functions in health and irritable bowel syndrome. Am J Physiol Gastrointest Liver Physiol. 2008 Aug;295(2):G219-25. doi: 10.1152/ajpgi.90202.2008. Epub 2008 May 29. PMID 18511740
- [Background] Cohen H, Buskila D, Neumann L, Ebstein RP. Confirmation of an association between fibromyalgia and serotonin transporter promoter region (5- HTTLPR) polymorphism, and relationship to anxiety-related personality traits. Arthritis Rheum. 2002 Mar;46(3):845-7. doi: 10.1002/art.10103. No abstract available. PMID 11920428
- [Background] Foster DC, Sazenski TM, Stodgell CJ. Impact of genetic variation in interleukin-1 receptor antagonist and melanocortin-1 receptor genes on vulvar vestibulitis syndrome. J Reprod Med. 2004 Jul;49(7):503-9. PMID 15305821
- [Background] Duerr RH, Taylor KD, Brant SR, Rioux JD, Silverberg MS, Daly MJ, Steinhart AH, Abraham C, Regueiro M, Griffiths A, Dassopoulos T, Bitton A, Yang H, Targan S, Datta LW, Kistner EO, Schumm LP, Lee AT, Gregersen PK, Barmada MM, Rotter JI, Nicolae DL, Cho JH. A genome-wide association study identifies IL23R as an inflammatory bowel disease gene. Science. 2006 Dec 1;314(5804):1461-3. doi: 10.1126/science.1135245. Epub 2006 Oct 26. PMID 17068223
- [Background] Tegeder I, Costigan M, Griffin RS, Abele A, Belfer I, Schmidt H, Ehnert C, Nejim J, Marian C, Scholz J, Wu T, Allchorne A, Diatchenko L, Binshtok AM, Goldman D, Adolph J, Sama S, Atlas SJ, Carlezon WA, Parsegian A, Lotsch J, Fillingim RB, Maixner W, Geisslinger G, Max MB, Woolf CJ. GTP cyclohydrolase and tetrahydrobiopterin regulate pain sensitivity and persistence. Nat Med. 2006 Nov;12(11):1269-77. doi: 10.1038/nm1490. Epub 2006 Oct 22. PMID 17057711
- [Background] Oertel B, Lotsch J. Genetic mutations that prevent pain: implications for future pain medication. Pharmacogenomics. 2008 Feb;9(2):179-94. doi: 10.2217/14622416.9.2.179. PMID 18370847
- [Background] De Vries B, Haan J, Frants RR, Van den Maagdenberg AM, Ferrari MD. Genetic biomarkers for migraine. Headache. 2006 Jul-Aug;46(7):1059-68. doi: 10.1111/j.1526-4610.2006.00499.x. PMID 16866710
- [Background] Reimann F, Cox JJ, Belfer I, Diatchenko L, Zaykin DV, McHale DP, Drenth JP, Dai F, Wheeler J, Sanders F, Wood L, Wu TX, Karppinen J, Nikolajsen L, Mannikko M, Max MB, Kiselycznyk C, Poddar M, Te Morsche RH, Smith S, Gibson D, Kelempisioti A, Maixner W, Gribble FM, Woods CG. Pain perception is altered by a nucleotide polymorphism in SCN9A. Proc Natl Acad Sci U S A. 2010 Mar 16;107(11):5148-53. doi: 10.1073/pnas.0913181107. Epub 2010 Mar 8. PMID 20212137
- [Background] Derogatis L. SCL-90-R Administration, Scoring and Procedures Manual-II. Clinical Psychometric Research Towson, MD, 1983:14-5.
- [Background] Taylor S, Zvolensky MJ, Cox BJ, Deacon B, Heimberg RG, Ledley DR, Abramowitz JS, Holaway RM, Sandin B, Stewart SH, Coles M, Eng W, Daly ES, Arrindell WA, Bouvard M, Cardenas SJ. Robust dimensions of anxiety sensitivity: development and initial validation of the Anxiety Sensitivity Index-3. Psychol Assess. 2007 Jun;19(2):176-88. doi: 10.1037/1040-3590.19.2.176. PMID 17563199
- [Background] Turk DC. A diathesis-stress model of chronic pain and disability following traumatic injury. Pain Res Manag. 2002 Spring;7(1):9-19. doi: 10.1155/2002/252904. PMID 16231063
- [Background] McCracken LM, Dhingra L. A short version of the Pain Anxiety Symptoms Scale (PASS-20): preliminary development and validity. Pain Res Manag. 2002 Spring;7(1):45-50. doi: 10.1155/2002/517163. PMID 16231066
- [Background] Leeuw M, Goossens ME, Linton SJ, Crombez G, Boersma K, Vlaeyen JW. The fear-avoidance model of musculoskeletal pain: current state of scientific evidence. J Behav Med. 2007 Feb;30(1):77-94. doi: 10.1007/s10865-006-9085-0. Epub 2006 Dec 20. PMID 17180640
- [Background] Sullivan M, Bishop S, Pivik J. The Pain Catastrophizing Scale: Development and Validation. . Psychological Assessment 1995;7:524-32.
- [Background] Katz J, Cohen L. Preventive analgesia is associated with reduced pain disability 3 weeks but not 6 months after major gynecologic surgery by laparotomy. Anesthesiology. 2004 Jul;101(1):169-74. doi: 10.1097/00000542-200407000-00026. PMID 15220787
- [Background] Costigan M, Scholz J, Woolf CJ. Neuropathic pain: a maladaptive response of the nervous system to damage. Annu Rev Neurosci. 2009;32:1-32. doi: 10.1146/annurev.neuro.051508.135531. PMID 19400724
- [Background] Birklein F, Riedl B, Neundorfer B, Handwerker HO. Sympathetic vasoconstrictor reflex pattern in patients with complex regional pain syndrome. Pain. 1998 Mar;75(1):93-100. doi: 10.1016/S0304-3959(97)00209-1. PMID 9539678
- [Background] Diatchenko L, Anderson AD, Slade GD, Fillingim RB, Shabalina SA, Higgins TJ, Sama S, Belfer I, Goldman D, Max MB, Weir BS, Maixner W. Three major haplotypes of the beta2 adrenergic receptor define psychological profile, blood pressure, and the risk for development of a common musculoskeletal pain disorder. Am J Med Genet B Neuropsychiatr Genet. 2006 Jul 5;141B(5):449-62. doi: 10.1002/ajmg.b.30324. PMID 16741943
- [Background] Modir JG, Wallace MS. Human experimental pain models 2: the cold pressor model. Methods Mol Biol. 2010;617:165-8. doi: 10.1007/978-1-60327-323-7_13. PMID 20336421
- [Background] Macrae WA. Chronic post-surgical pain: 10 years on. Br J Anaesth. 2008 Jul;101(1):77-86. doi: 10.1093/bja/aen099. Epub 2008 Apr 22. PMID 18434337
- [Background] Edwards CL, Fillingim RB, Keefe F. Race, ethnicity and pain. Pain. 2001 Nov;94(2):133-137. doi: 10.1016/S0304-3959(01)00408-0. PMID 11690726
- [Background] Katz J, Melzack R. Measurement of pain. Surg Clin North Am. 1999 Apr;79(2):231-52. doi: 10.1016/s0039-6109(05)70381-9. PMID 10352653
- [Background] Dworkin RH, Turk DC, Revicki DA, Harding G, Coyne KS, Peirce-Sandner S, Bhagwat D, Everton D, Burke LB, Cowan P, Farrar JT, Hertz S, Max MB, Rappaport BA, Melzack R. Development and initial validation of an expanded and revised version of the Short-form McGill Pain Questionnaire (SF-MPQ-2). Pain. 2009 Jul;144(1-2):35-42. doi: 10.1016/j.pain.2009.02.007. Epub 2009 Apr 7. PMID 19356853
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Bennett MI, Smith BH, Torrance N, Potter J. The S-LANSS score for identifying pain of predominantly neuropathic origin: validation for use in clinical and postal research. J Pain. 2005 Mar;6(3):149-58. doi: 10.1016/j.jpain.2004.11.007. PMID 15772908
- [Background] Reiss S, Peterson RA, Gursky DM, McNally RJ. Anxiety sensitivity, anxiety frequency and the prediction of fearfulness. Behav Res Ther. 1986;24(1):1-8. doi: 10.1016/0005-7967(86)90143-9. No abstract available. PMID 3947307
- [Background] McCracken LM, Zayfert C, Gross RT. The Pain Anxiety Symptoms Scale: development and validation of a scale to measure fear of pain. Pain. 1992 Jul;50(1):67-73. doi: 10.1016/0304-3959(92)90113-P. PMID 1513605
- [Background] Pollard CA. Preliminary validity study of the pain disability index. Percept Mot Skills. 1984 Dec;59(3):974. doi: 10.2466/pms.1984.59.3.974. No abstract available. PMID 6240632
- [Background] Tait RC, Pollard CA, Margolis RB, Duckro PN, Krause SJ. The Pain Disability Index: psychometric and validity data. Arch Phys Med Rehabil. 1987 Jul;68(7):438-41. PMID 3606368
- [Background] Weathers F, Litz B, Huska J, Keane T. PCL-C for DSM-IV Boston: National Center for PTSD - Behavioral Science Division 1994.
- [Background] Blanchard EB, Jones-Alexander J, Buckley TC, Forneris CA. Psychometric properties of the PTSD Checklist (PCL). Behav Res Ther. 1996 Aug;34(8):669-73. doi: 10.1016/0005-7967(96)00033-2. PMID 8870294
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] McCracken LM, Vowles KE, Eccleston C. Acceptance of chronic pain: component analysis and a revised assessment method. Pain. 2004 Jan;107(1-2):159-66. doi: 10.1016/j.pain.2003.10.012. PMID 14715402
- [Background] Vowles KE, McCracken LM, McLeod C, Eccleston C. The Chronic Pain Acceptance Questionnaire: confirmatory factor analysis and identification of patient subgroups. Pain. 2008 Nov 30;140(2):284-291. doi: 10.1016/j.pain.2008.08.012. Epub 2008 Sep 27. PMID 18824301
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Carlson LE, Brown KW. Validation of the Mindful Attention Awareness Scale in a cancer population. J Psychosom Res. 2005 Jan;58(1):29-33. doi: 10.1016/j.jpsychores.2004.04.366. PMID 15771867
- [Background] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Background] Roosen K, Page MG, Kleiman V, Katz J. Sensitivity to pain traumatization scale (SPTS): Examining differences accross gender, pain history, and pain sensitivity. World Congress on Pain. Montreal, QC., 2010.
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cole RJ, Kripke DF, Gruen W, Mullaney DJ, Gillin JC. Automatic sleep/wake identification from wrist activity. Sleep. 1992 Oct;15(5):461-9. doi: 10.1093/sleep/15.5.461. PMID 1455130
- [Background] Lichstein KL, Stone KC, Donaldson J, Nau SD, Soeffing JP, Murray D, Lester KW, Aguillard RN. Actigraphy validation with insomnia. Sleep. 2006 Feb;29(2):232-9. PMID 16494091
- [Background] Rolke R, Baron R, Maier C, Tolle TR, Treede -DR, Beyer A, Binder A, Birbaumer N, Birklein F, Botefur IC, Braune S, Flor H, Huge V, Klug R, Landwehrmeyer GB, Magerl W, Maihofner C, Rolko C, Schaub C, Scherens A, Sprenger T, Valet M, Wasserka B. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. Pain. 2006 Aug;123(3):231-243. doi: 10.1016/j.pain.2006.01.041. Epub 2006 May 11. PMID 16697110
- [Background] Bouhassira D, Kern D, Rouaud J, Pelle-Lancien E, Morain F. Investigation of the paradoxical painful sensation ('illusion of pain') produced by a thermal grill. Pain. 2005 Mar;114(1-2):160-7. doi: 10.1016/j.pain.2004.12.014. Epub 2005 Jan 20. PMID 15733641
- [Background] Craig BAD. Can the basis for central neuropathic pain be identified by using a thermal grill? Pain. 2008 Apr;135(3):215-216. doi: 10.1016/j.pain.2008.01.022. Epub 2008 Feb 20. No abstract available. PMID 18282660
- [Background] Rosa C, Ghione S, Mezzasalma L, Pellegrini M, Basile Fasolo C, Giaconi S, Gazzetti P, Ferdeghini M. Relationship between pain sensitivity, cardiovascular reactivity to cold pressor test and indexes of activity of the adrenergic and opioid system. Clin Exp Hypertens A. 1988;10 Suppl 1:383-90. doi: 10.3109/10641968809075994. PMID 3072126
- [Background] Coffman DL, MacCallum RC. Using Parcels to Convert Path Analysis Models Into Latent Variable Models. Multivariate Behav Res. 2005 Apr 1;40(2):235-59. doi: 10.1207/s15327906mbr4002_4. PMID 26760108
- [Background] Kline R. Principles and practice of structural equation modeling. 2nd ed. New York, NY: Guilford Press; 2005.
- [Background] Byrne B. Structural equation modeling with amos: Basic concepts, applications, and programming. Mahwah, NJ: Lawrence Erlbaum Associates; 2001.
- [Background] Maixner W, Diatchenko L, Fillingim RB, Greenspan J, Orbach R, Slade GD, Smith S. Assessment of biopsychosocial and genetic risk factors for chronic orofacial pain: the OPPERA Study. American Pain Society Meeting. Baltimore, Maryland, 2010.
- [Background] Storey JD, Tibshirani R. Statistical significance for genomewide studies. Proc Natl Acad Sci U S A. 2003 Aug 5;100(16):9440-5. doi: 10.1073/pnas.1530509100. Epub 2003 Jul 25. PMID 12883005
- [Derived] Xiao MZX, Khan JS, Dana E, Rao V, Djaiani G, Richebe P, Katz J, Wong D, Clarke H. Prevalence and Risk Factors for Chronic Postsurgical Pain after Cardiac Surgery: A Single-center Prospective Cohort Study. Anesthesiology. 2023 Sep 1;139(3):309-320. doi: 10.1097/ALN.0000000000004621. PMID 37192204